CLINICAL TRIAL: NCT05232929
Title: Long-term Follow-up Study of Patients With Spinal Muscular Atrophy Receiving Risdiplam Treatment
Brief Title: Long-term Follow-up Study of Risdiplam in Participants With Spinal Muscular Atrophy (SMA)
Acronym: WeSMA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML43702
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Risdiplam (Experimental): Participants who are taking risdiplam prescribed based on clinician judgment, as per the Evrysdi® USPI are enrolled in this study.
  A Remote Virtual Site option is available in the study allowing enrollment of participants with SMA who are prescribed risdiplam treatment even if their physician is not a participating investigator. A central investigator will be responsible for data collection and data entry for participants who do not have a participating investigator.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Risdiplam taken by participants as prescribed by their physician.
  Other Names: Evrysdi®

SUMMARY:
A multi-center, longitudinal, prospective, non-comparative study to investigate the long-term safety and effectiveness of risdiplam, prescribed based on clinician judgment as per the Evrysdi® U.S. Package Information (USPI) in adult and pediatric participants with SMA. In this study, participants will be followed for approximately 24 months from enrollment or until withdrawal of consent, loss to follow-up, or death. Participants who discontinue risdiplam may still remain in the study if they agree to continue participating in the follow-up assessments.

An optional sub-study was planned to assess the feasibility, acceptability, and adherence of remote assessment of motor and bulbar functions in participants with SMA using wearable and smartphone-based biosensors. This substudy was withdrawn upon implementation of protocol version 4.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent or assent when appropriate, as determined by the participant's age and individual site and local standards
* Prescribed or continued risdiplam based on clinical judgment of prescriber, as per the risdiplam (Evrysdi) USPI, after U.S. FDA approval (07 August 2020)

Exclusion Criteria:

* Hypersensitivity to risdiplam
* Participated in a registrational trial for risdiplam (i.e., Firefish [NCT02913482], Sunfish [NCT02908685], Jewelfish [NCT03032172], and Rainbowfish [NCT03779334])

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) | From enrollment up to the duration of the study or until withdrawal of consent, loss to follow-up, or death (up to approximately 24 months)
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as AE.

SECONDARY OUTCOMES:
Percentage of Participants Considered Improved on the Clinical Global Impression of Change (CGI-C) Scale | From enrollment up to the duration of the study or until withdrawal of consent, loss to follow-up, or death (up to approximately 24 months)
  The CGI-C is used to score a clinician's impression of a participant's change in global health. The CGI-C is a single item measure of change in global health, using seven response options: "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", and "very much worse". Participants considered as "improved" include responses of "very much improved, "much improved" and "minimally improved".

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (37):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Health Care, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - University California - Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Hospital, Washington D.C., District of Columbia
  - Nemour's Children's Hospital, Florida, Orlando, Florida
  - All Children's Research Institute, Inc., St. Petersburg, Florida
  - Advent Health Orlando, Winter Park, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Pediatric Rehabilitation Center, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Gillette Children's Specialty Healthcare, Minnetonka, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University;Wash Uni. Sch. Of Med, St Louis, Missouri
  - NYU Hospital for Joint Diseases, New York, New York
  - Columbia University Med Center, New York, New York
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas at Austin Health sciences, Dell Medical School, Austin, Texas
  - Neurology & Neuromuscular Care Center, Denton, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University Of Utah, Salt Lake City, Utah
  - University of Virginia Children?s Hospital, Charlottesville, Virginia
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - UBC (Remote Coordinating Center, no physical facility), Morgantown, West Virginia
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Instituto de Rehabilitación del Caribe, Santurce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing